CLINICAL TRIAL: NCT00410423
Title: Phase I/II Trial of VELCADE® (Bortezomib) in Combination With Mitoxantrone and Etoposide for Relapsed or Refractory Acute Leukemias
Brief Title: Study of VELCADE® With Mitoxantrone and Etoposide for Leukemias
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06U.70; 2005-74 (Other: CCRRC); JT 1162 (Other: JeffTrial Number)
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Relapsed Acute Leukemia; Refractory Acute Leukemia
Keywords: Leukemia; Acute Myeloid Leukemia; Acute Lymphoid / Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Bortezomib; Mitoxantrone; Etoposide; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bortezomib 0.7mg/m^2 (Experimental): Bortezomib in combination with mitoxantrone, etoposide and cytarabine
  Interventions: Drug: Bortezomib with mitoxantrone, etoposide and cytarabine
- Bortezomib 1.0mg/m^2 (Experimental)
  Interventions: Drug: Bortezomib 1.0mg/m^2
- Bortezomib 1.3mg/m^2 (Experimental)
  Interventions: Drug: Bortezomib 1.3mg/m^2

INTERVENTIONS:
Drug: Bortezomib with mitoxantrone, etoposide and cytarabine — All patients receive bortezomib in combination with mitoxantrone, etoposide and cytarabine. This is a 5 day chemotherapy regimen that is administered in the hospital.
  Other Names: Velcade
  Arms: Bortezomib 0.7mg/m^2
Drug: Bortezomib 1.0mg/m^2 — All patients receive bortezomib in combination with mitoxantrone, etoposide and cytarabine. This is a 5 day chemotherapy regimen that is administered in the hospital.
  Other Names: Velcade
  Arms: Bortezomib 1.0mg/m^2
Drug: Bortezomib 1.3mg/m^2 — All patients receive bortezomib in combination with mitoxantrone, etoposide and cytarabine. This is a 5 day chemotherapy regimen that is administered in the hospital.
  Other Names: Velcade
  Arms: Bortezomib 1.3mg/m^2

SUMMARY:
Based on what is known about it's mechanism of action, bortezomib is presumed to make other chemotherapy drugs work better. This study examines the use of bortezomib in combination with an already effective chemotherapy regimen that is used to treat leukemias that have relapsed or been refractory to treatment.

DETAILED DESCRIPTION:
VELCADE is a drug that blocks growth of cancer cells and helps destroy them. This research will help us to determine if VELCADE when combined with chemotherapy is useful in treating the leukemia with which you have been diagnosed. Your leukemia is a type that did not respond to chemotherapy or has come back after successful therapy.

VELCADE is approved by the Food and Drug Administration (FDA) for the treatment of multiple myeloma for patients that have received at least one prior therapy. Multiple Myeloma is a type of cancer that develops from blood cells. The dose of the drug being used in this research study is the same as what is used for the treatment of myeloma but the number of injections is less. VELCADE has, however not been approved by the FDA for use in acute leukemia. Mitoxantrone and etoposide, the other two chemotherapy drugs are also used for treating leukemia.

In the first part of the study, we are going to test the safety of VELCADE at different doses when given with mitoxantrone and etoposide. You may be enrolled at any one of three doses. In the second part, we are going to assess the response to the combination of VELCADE and chemotherapy drugs. You will receive VELCADE at the chosen dose based on safety assessment from Phase I. It will be administered as an intravenous (through the vein) injection on day-1 and day-4 of the 5-day schedule. In addition, you will also receive mitoxantrone over 15 minutes and etoposide over 45 minutes from days 1-5. The first 28 days from the beginning of the treatment will be called a treatment cycle.

On day-14 of the treatment cycle, you will have a bone marrow biopsy done to see if all the leukemia cells have disappeared. If there is no evidence of leukemia, then you may receive growth factors to help your marrow recover faster. If there is still presence of leukemia, in the same amount or more, then the treatment will be considered a failure and you will not receive any more of this treatment.

If there is a partial improvement then you will receive additional cycles of VELCADE with chemotherapy as described above until there are no signs of your disease. This is called a complete remission.

Therapy will be withheld at any time if there is concern that you are having side-effects that are not medically acceptable. Once the side-effects have resolved, VELCADE therapy may be re-started at a lower dose.

It is estimated that you may require about two to three cycles of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (ie, a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male subject agrees to use an acceptable method for contraception for the duration of the study.
* Patients who have had a diagnosis of Acute Myeloid Leukemia (AML) or Acute Lymphoblastic Leukemia (ALL) will be eligible for the study.

  * Patients must have failed initial therapy that may manifest in either of the following ways:

    * Demonstration of Primary Refractory Disease (Primary Induction Failure) as evidenced by a mid-cycle bone marrow analysis showing lack of complete tumor clearance (CTC).
    * Relapse of initial disease after a period of attaining complete remission.
* Patients must be > 18 years of age, with no upper age limit.
* ECOG performance status of 0 or 1.
* Patients have no symptomatic cardiac or pulmonary disease and adequate hepatic and renal function as measured by the following criteria:

  * Cardiac: Left ventricular ejection fraction at rest must be >40% (MUGA preferred)
  * Hepatic: ALT and AST < 3x the upper limits of normal range as specified by the institution's clinical laboratory.
  * Renal: Serum creatinine within the normal range (< 1.4 mg/dL) or if creatinine outside normal range then creatinine clearance > 60 mL/min/m2
* Patients who have had a diagnosis of Acute Myeloid Leukemia (AML) or Acute Lymphoblastic Leukemia (ALL) will be eligible for the study.
* Patients must have failed initial therapy that may manifest in either of the following ways:

  * Demonstration of Primary Refractory Disease (Primary Induction Failure) as evidenced by a mid-cycle bone marrow analysis showing lack of complete tumor clearance (CTC).
  * Relapse of initial disease after a period of attaining complete remission.
* Patients must be > 18 years of age, with no upper age limit.
* ECOG performance status of 0 or 1.
* Patients have no symptomatic cardiac or pulmonary disease and adequate hepatic and renal function as measured by the following criteria:

  * Cardiac: Left ventricular ejection fraction at rest must be >40% (MUGA preferred)
  * Hepatic: ALT and AST < 3x the upper limits of normal range as specified by the institution's clinical laboratory.
  * Renal: Serum creatinine within the normal range (< 1.4 mg/dL) or if creatinine outside normal range then creatinine clearance > 60 mL/min/m2

Exclusion Criteria:

* Patient has > Grade 2 peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has New York Hospital Association (NYHA) Class III or IV heart failure (see section 8.4), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to bortezomib, boron or mannitol.
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum or urinary pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has received other investigational drugs within 14 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-01; Primary Completion 2013-05 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Filicko-O'Hara, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 - Bortezomib 0.7mg/m^2; Phase 1 - Bortezomib 1.0 mg/m^2; Phase 1 - Bortezomib 1.3 mg/m^2; Phase 2 - Bortezomib 1.3mg/m^2: Bortezomib in combination with mitoxantrone, etoposide and cytarabine
  Bortezomib with mitoxantrone, etoposide and cytarabine: All patients receive bortezomib in combination with mitoxantrone, etoposide and cytarabine. This is a 5 day chemotherapy regimen that is administered in the hospital.
Period: Phase 1 - Dose Level 1
Arm/Group | Phase 1 - Bortezomib 0.7mg/m^2 | Phase 1 - Bortezomib 1.0 mg/m^2 | Phase 1 - Bortezomib 1.3 mg/m^2 | Phase 2 - Bortezomib 1.3mg/m^2
Started | 3 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Phase 1 - Dose Level 2
Arm/Group | Phase 1 - Bortezomib 0.7mg/m^2 | Phase 1 - Bortezomib 1.0 mg/m^2 | Phase 1 - Bortezomib 1.3 mg/m^2 | Phase 2 - Bortezomib 1.3mg/m^2
Started | 0 | 5 | 0 | 0
Completed | 0 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Phase 1 - Dose Level 3
Arm/Group | Phase 1 - Bortezomib 0.7mg/m^2 | Phase 1 - Bortezomib 1.0 mg/m^2 | Phase 1 - Bortezomib 1.3 mg/m^2 | Phase 2 - Bortezomib 1.3mg/m^2
Started | 0 | 0 | 3 | 0
Completed | 0 | 0 | 3 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1 - Bortezomib 0.7mg/m^2 | Phase 1 - Bortezomib 1.0 mg/m^2 | Phase 1 - Bortezomib 1.3 mg/m^2 | Phase 2 - Bortezomib 1.3mg/m^2
Started | 0 | 0 | 0 | 44
Completed | 0 | 0 | 0 | 44
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Bortezomib: Bortezomib in combination with mitoxantrone, etoposide and cytarabine
  Bortezomib with mitoxantrone, etoposide and cytarabine: All patients receive bortezomib in combination with mitoxantrone, etoposide and cytarabine. This is a 5 day chemotherapy regimen that is administered in the hospital.
Arm/Group | Bortezomib
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.39 (15.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 35
  More than one race | 0
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity in Phase I
Description: Dose limiting toxicity (DLT) is defined as grade-3 toxicity definitely related to bortezomib or grade-4 toxicity probably or definitely related to bortezomib.
Time Frame: 30-90 days
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 - Bortezomib 1.3mg/m^2: Bortezomib in combination with mitoxantrone, etoposide and cytarabine
  Bortezomib with mitoxantrone, etoposide and cytarabine: All patients receive bortezomib in combination with mitoxantrone, etoposide and cytarabine. This is a 5 day chemotherapy regimen that is administered in the hospital.
Arm/Group | Phase 1 - Bortezomib 0.7mg/m^2 | Phase 1 - Bortezomib 1.0 mg/m^2 | Phase 1 - Bortezomib 1.3mg/m^2
Number analyzed (Participants) | 3 | 5 | 3
Participants | 0 | 0 | 0

2. Primary Outcome: Complete Response Rate to 1.3mg/m^2 of Bortezomib With Mitoxantrone and Etoposide in Phase II
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions.
  The percentage of participants that experienced complete response will be reported.
Time Frame: Up to 7 years
Measure: Number; unit: percentage of participants
Groups:
- Phase 2 - Bortezomib 1.3mg/m^2: Bortezomib 1.3mg/m2: All patients receive bortezomib in combination with mitoxantrone, etoposide and cytarabine. This is a 5 day chemotherapy regimen that is administered in the hospital.
Arm/Group | Phase 2 - Bortezomib 1.3mg/m^2
Number analyzed (Participants) | 44
percentage of participants | 27

ADVERSE EVENTS:
Description: Adverse events not available for 17 patients--these patients are excluded from adverse event counts
Arm/Group | Bortezomib
Serious Adverse Events (participants affected / at risk) | 10/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib (N=38)
Cough (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (9)
Infection (Infections and infestations) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib (N=38)
Abdominal pain (General disorders) | 10 (11)
Achiness (General disorders) | 2 (2)
Acute infusion reaction (General disorders) | 7 (13)
Allergic reaction (General disorders) | 3 (7)
Alopecia (General disorders) | 6 (6)
Anorexia (General disorders) | 16 (19)
Anxiety (Psychiatric disorders) | 8 (8)
Arm pain (General disorders) | 3 (4)
Ataxia (Nervous system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Back pain (General disorders) | 7 (8)
Bladder stone (Renal and urinary disorders) | 1 (1)
Bleeding (Blood and lymphatic system disorders) | 3 (4)
Bloating (Gastrointestinal disorders) | 2 (2)
Blood-tinged mucus (General disorders) | 1 (1)
Bone pain (General disorders) | 3 (4)
Breast mass (General disorders) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 3 (3)
Bump on finger (General disorders) | 1 (1)
Calf pain (General disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 2 (2)
Change in vision (Eye disorders) | 3 (3)
Chest pain (General disorders) | 6 (7)
Chills (General disorders) | 10 (11)
Chronic rhinsinusitis (General disorders) | 1 (1)
Clostridium difficile (Infections and infestations) | 1 (1)
Congestive heart failure (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 14 (17)
Cough (General disorders) | 9 (10)
Decreased appetite (General disorders) | 3 (3)
Dehydration (General disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 19 (19)
Distended abdomen (Gastrointestinal disorders) | 3 (3)
Dizziness (General disorders) | 9 (9)
Dry cough (General disorders) | 1 (1)
Dry eyes (Eye disorders) | 1 (1)
Dry mouth (General disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dry, cracked lips (General disorders) | 2 (2)
Dysgeusia (General disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (General disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (12)
Dysuria (Renal and urinary disorders) | 1 (2)
Edema (Skin and subcutaneous tissue disorders) | 18 (21)
Elbow pain (General disorders) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1)
Epistaxis (General disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Facial swelling (General disorders) | 1 (1)
Fatigue (General disorders) | 18 (19)
Febrile neutropenia (Blood and lymphatic system disorders) | 12 (14)
Fever (General disorders) | 9 (12)
Fistula (General disorders) | 1 (1)
Flank pain (General disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Fluid retention (General disorders) | 1 (1)
Flushing (Skin and subcutaneous tissue disorders) | 2 (2)
Foot pain (General disorders) | 1 (1)
Gas pain (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Genitourinary obstruction (Renal and urinary disorders) | 1 (1)
Gum swelling (General disorders) | 1 (1)
Hand pain (General disorders) | 2 (2)
Headache (General disorders) | 17 (19)
Heartburn (Gastrointestinal disorders) | 1 (1)
Hematuria (Blood and lymphatic system disorders) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 4 (4)
Hives (Skin and subcutaneous tissue disorders) | 3 (3)
Hoarseness (General disorders) | 1 (1)
Hot flashes (General disorders) | 1 (1)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 2 (2)
Hyperkalemia (Blood and lymphatic system disorders) | 1 (1)
Hyperphosphatemia (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Blood and lymphatic system disorders) | 6 (6)
Hyperuricemia (Blood and lymphatic system disorders) | 1 (1)
Hypoglycemia (Blood and lymphatic system disorders) | 2 (2)
Hypokalemia (Blood and lymphatic system disorders) | 5 (5)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1)
Hypophosphatemia (Blood and lymphatic system disorders) | 1 (1)
Hypotension (Blood and lymphatic system disorders) | 16 (18)
Hypothyroidism (Endocrine disorders) | 1 (1)
Incontinence of stool (General disorders) | 1 (1)
Increased alklaline phosphatase (Blood and lymphatic system disorders) | 2 (2)
Increased ALT (Blood and lymphatic system disorders) | 3 (6)
Increased AST (Blood and lymphatic system disorders) | 3 (3)
Increased creatinine (Blood and lymphatic system disorders) | 1 (1)
Infection (Infections and infestations) | 3 (3)
Insomnia (General disorders) | 5 (5)
Iron overload (General disorders) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 5 (5)
Itchy eyes (Eye disorders) | 1 (1)
Joint pain (General disorders) | 2 (2)
Knee pain (General disorders) | 1 (1)
Leg pain (General disorders) | 4 (5)
Lesion (Skin and subcutaneous tissue disorders) | 2 (2)
Liver dysfunction (Hepatobiliary disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 16 (17)
Muscle cramping (General disorders) | 1 (1)
Muscle pain (General disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nausea (General disorders) | 27 (32)
Neck pain (General disorders) | 3 (3)
Neuropathy (Nervous system disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Night sweats (General disorders) | 1 (1)
Oral pain (General disorders) | 4 (4)
Oral thrush (General disorders) | 3 (3)
Pain at femoral line site (General disorders) | 1 (1)
Pain at PICC site (General disorders) | 5 (5)
Pain from bone marrow biopsy (General disorders) | 6 (6)
Pain from mouth sore (General disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 15 (16)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis (General disorders) | 2 (3)
Rib pain (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Shoulder pain (General disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus congestion (General disorders) | 1 (1)
Sinus headache (General disorders) | 2 (2)
Sinus pain (General disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 7 (7)
Sinusitis (General disorders) | 3 (3)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Sore in mouth (General disorders) | 2 (3)
Sore throat (General disorders) | 3 (3)
Sternal pain (General disorders) | 1 (1)
Stomach pain (General disorders) | 1 (1)
Strong urine odor (Renal and urinary disorders) | 1 (1)
Sweating (General disorders) | 4 (4)
Swelling of parotid gland (General disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 8 (8)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thigh pain (General disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Tingling in fingertips (Nervous system disorders) | 1 (1)
Tingling in palms (Nervous system disorders) | 1 (1)
Toe pain (General disorders) | 1 (1)
Tongue pain (General disorders) | 1 (1)
Tooth pain (General disorders) | 1 (1)
Tremors (General disorders) | 2 (2)
Trouble sleeping (General disorders) | 2 (2)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 5 (5)
Urinary retention (Renal and urinary disorders) | 3 (3)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Weakness (General disorders) | 13 (13)
Weight gain (General disorders) | 1 (2)
Weight loss (General disorders) | 1 (1)
Wheezing (General disorders) | 1 (1)
Lethargy (General disorders) | 1 (1)
Tingling in toes (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes